CLINICAL TRIAL: NCT03953014
Title: Pharmacogenetics of Antidepressant-Induced Disinhibition in Children Study
Brief Title: Pharmacogenetics of Antidepressant-Induced Disinhibition
Acronym: PGx-AID
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Other Study IDs: REB18-0519
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Obsessive-Compulsive Disorder; Anxiety Disorders; Major Depressive Disorder; Antidepressant Drug Adverse Reaction
Keywords: SSRI; Depression; Children; OCD; Anxiety; Antidepressants
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — We will be collecting a 4mL saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify pharmacogenetic profiles associated with selective serotonin reuptake inhibitors (SSRI)-induced behavioral disinhibition in children with Major depressive disorder (MDD), anxiety disorders and/or obsessive-compulsive disorder (OCD) that could be used clinically to reduce the incidence of this adverse event and improve health outcomes.

DETAILED DESCRIPTION:
Background and Rationale:

Antidepressants such as serotonin-selective reuptake inhibitors (SSRIs) are frequently prescribed to children to manage major depressive and anxiety disorders. Although SSRIs are thought to be generally effective and well-tolerated in children, 10%- 20% of children treated with SSRIs experience behavioral disinhibition (i.e. activation, hyperactivity, impulsivity, insomnia) that can lead to devastating consequences (e.g. suicidal impulses, violence). There are currently no tools available to assist healthcare providers in predicting which children will experience behavioral disinhibition as a result of SSRI treatment.

Research Question:

Do children who experience SSRI-induced behavioral disinhibition (SIBD) have a distinct pharmacogenetic profile relative to children who do not have these adverse experiences?

Methodology:

Using a retrospective cohort study design, 120 SSRI-treated children diagnose with major depression, anxiety and OCD, aged 6 to 17 years of aged will be recruited from Child and Adolescent Addiction, Mental Health & Psychiatry (CAAMHP) Program in Calgary. Children with a current or past history of SSRI use will be identified via recruitment advertisements and by CAAMHP treatment teams operating within community clinics as well as inpatient units within the Alberta Children's Hospital and Foothills Medical Centre.

Clinical data will be collected from the participant's medical record as well as information provided by the child's healthcare provider and caretaker using a customized data collection form. Saliva will be collected, processed and genotyped in accordance with standard procedures. Participants and their parents will complete self-report measures to gather information regarding demographics, SIBD, and other adverse side effects and drug reactions.

Using machine learning (i.e. the construction of algorithms that can learn from and make predictions on data) we will identify and validate a panel of genetic variants that could be used to pre-emptively detect children at-risk for developing SSRI-induced behavioral disinhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 - 24 years
2. Medical records available
3. Diagnosis of MDD, anxiety disorder, or OCD
4. Current or past history of SSRI therapy

Exclusion Criteria:

1. Inability of parent/legal guardian to give informed consent
2. Inability of the child to give informed assent
3. Unwillingness of child to provide saliva sample for genetic analysis
4. Current, past or suspected diagnosis of attention deficit hyperactivity disorder, oppositional defiant disorder, conduct disorder, bipolar disorder, psychotic disorder, or pervasive developmental disorder.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: SSRI-treated children diagnosed with major depression, anxiety and OCD, aged 6 to 24 years recruited from the Child and Adolescent Addiction, Mental Health & Psychiatry (CAAMP) Program in Calgary.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Genetic variants in SSRI metabolism | 4 years
  DNA Sample Collection & Genotyping. Saliva will be collected using Oragene® collection tubes (DNA Genotek, Ottawa, Canada). DNA will be extracted using standard procedures and genotyped.
Behavioural Disinhibition | 4 years
  Information on behavioural disinhibition (BD) to note the type, duration and severity of BD gathered from medical records, and participant and parent report.
  The Treatment-emergent activation and suicidality assessment profile (TEASAP), is a questionnaire that assess common symptoms of activation syndrome/behavioural disinhibition in youth due to SSRI usage.

SECONDARY OUTCOMES:
Adverse Drug Reactions other than SIBD | 4 years
  A self-report instrument, The Antidepressant Side-Effect Checklist (ASEC) will be used to assess the presence of common adverse reactions to antidepressants.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Bousman, PhD, Principal Investigator — University of Calgary; Paul Arnold, MD, Principal Investigator — University of Calgary
Locations (1):
- Child and Adolescent Addiction, Mental Health & Psychiatry, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No